CLINICAL TRIAL: NCT00549068
Title: Impact of NTx Point of Care (POC) Device on Patient Satisfication With Actonel 35mg Once a Seek Treatment a Multicenter Prospective Open Label Randomized Controlled Community Practice-based Study
Brief Title: POWER Point of Care Effect on Satisfaction of Treatment
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Sanofi (Industry)
Collaborators: Procter and Gamble (Industry)
Responsible Party: Study Director, sanofi-aventis
Allocation: Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: HMR4003B_4031
Record Dates: First submitted 2007-10-24; First posted 2007-10-25 (Estimated); Last update posted 2009-12-07 (Estimated); Status verified 2009-12

CONDITIONS: Osteoporosis, Postmenopausal
MeSH Terms: conditions — Osteoporosis, Postmenopausal | interventions — Risedronic Acid

INTERVENTIONS:
Drug: Risedronate Sodium (Actonel)

SUMMARY:
To compare the subject satisfaction rating in women treated for postmenopausal osteoporosis with Actonel 35mg Once-a-Week for 24 weeks, and receiving feedback information, after 12 weeks of treatment, based on bone resorption marker results using the NTx Point-Of-Care (POC) device, to similar women treated as per regular clinical practice

ELIGIBILITY:
Inclusion Criteria:

* Women diagnosed with postmenopausal osteoporosis using community practice standards
* Women previously non-treated for osteoporosis, OR treated for osteoporosis with biphosphonates (alendronate, etidronate), hormone replacement therapy estrogen, estrogen-related drugs, progesterone, subcutaneous estrogen implant), raloxifene, fluoride, or calcitonin within the past 2 years but discontinued prior to enrolment into the study either due to:lack of effect or intolerance

Exclusion Criteria:

* Subjects treated with Actonelr 5 mg daily,
* Mental condition rendering the subject unable to understand the nature, scope, and possible consequences of the study
* Subject unlikely to comply with protocol, e.g., uncooperative attitude, inability to return for follow-up visits, and unlikelihood of completing the study
* Known/Suspected hypersensitivity to any component of Actonelr 35 mg Once-a-Week
* Known/Suspected hypocalcaemia
* Known/Suspected severe renal impairment (creatinine clearance < 30ml/min)
* Known/Suspected hyperparathyroidism
* Known/Suspected hyperthyroidism
* Known/Suspected active urinary tract infection
* Known high urine levels of calcium (3 4mg/ml)

The above information is not intended to contain all considerations relevant to a patient's potential participation in a clinical trial.

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 2433 (Actual)
Dates: Start 2003-02; Study Completion 2004-11 (Actual)

PRIMARY OUTCOMES:
Compare subject satisfaction rating in women treated for postmenopausal osteoporosis with Actonel® 35 mg Once-a-Week for 24 weeks, and receiving feedback information after 12 weeks of treatment to similar women monitored as per regular clinical practice

SECONDARY OUTCOMES:
Compare subject satisfaction with Actonel® 35 mg Once-a-Week in subject subgroups: previously treated with biphosphonates, HRT, raloxifene, fluoride, or calcitonin within past 2 years vs. those previously non treated

CONTACTS AND LOCATIONS:
Overall Officials: Mary Tzortzis, Study Director — Sanofi